CLINICAL TRIAL: NCT03443947
Title: Modified Mallampati Scoring Technique for Airway Assessment
Acronym: mod mallampati
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: AlRefaey Kandeel (Other)
Responsible Party: Sponsor-Investigator, AlRefaey Kandeel, lecturer, Mansoura University
Organization: Mansoura University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Dr Waleed 1
Record Dates: First submitted 2018-01-03; First posted 2018-02-23 (Actual); Last update posted 2018-02-23 (Actual); Status verified 2018-02

CONDITIONS: Intubation;Difficult
MeSH Terms: interventions — Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- D group (Experimental)
  Interventions: Device: Tongue depressor group; Procedure: control group

INTERVENTIONS:
Device: Tongue depressor group — using a tongue depressor to assess airway score without tongue protrusion
Procedure: control group — airway assessment after tongue protrusion

SUMMARY:
comparing a new technique for airway assessment using tongue depressor versus conventional mallampati scoring system. Using tongue depressor to improve airway score is suggested to increase reliability of airway assessment model

ELIGIBILITY:
Inclusion Criteria:

* all patients scheduled for elective surgery

Exclusion Criteria:

* known difficult airway trismus cases maxillofacial anomalies

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2018-03-01 (Estimated); Primary Completion 2018-12-31 (Estimated); Study Completion 2018-12-31 (Estimated)

PRIMARY OUTCOMES:
assessment of airway difficulty | before intubation
  correlation between airway score and view during laryngoscopy

CONTACTS AND LOCATIONS:
Locations (2):
- Egypt (2):
  - Mansoura university, Al Manşūrah, Dkahleya
  - Gastroenterology center, Al Mansurah

IPD SHARING:
Plan to Share IPD: Undecided